CLINICAL TRIAL: NCT03175120
Title: A Trial Comparing the Efficacy and Safety of Insulin Degludec/Liraglutide and Insulin Degludec in Combination With Metformin in Chinese Subjects With Type 2 Diabetes Mellitus Inadequately Controlled With Basal Insulin Therapy and Metformin With or Without One Other OAD
Brief Title: A Trial Comparing Insulin Degludec/Liraglutide and Insulin Degludec in Combination With Metformin in Chinese Subjects With Type 2 Diabetes Mellitus Inadequately Controlled With Basal Insulin Therapy and Metformin With or Without One Other Oral Antidiabetic Drug (OAD)
Acronym: DUAL™ II China
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN9068-4166; U1111-1154-6732 (Other: World Health Organization (WHO)); CTR20060909 (Registry Identifier: China Drug Trials (China))
Record Dates: First submitted 2017-05-24; First posted 2017-06-05 (Actual); Results first posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — IDegLira; insulin degludec

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Insulin degludec/liraglutide (Experimental)
  Interventions: Drug: Insulin degludec/liraglutide
- Insulin degludec (Active Comparator)
  Interventions: Drug: Insulin degludec

INTERVENTIONS:
Drug: Insulin degludec/liraglutide — Administered subcutaneously (s.c., under the skin) once daily in combination with metformin for the treatment duration of 26 weeks.
  Arms: Insulin degludec/liraglutide
Drug: Insulin degludec — Administered subcutaneously (s.c., under the skin) once daily in combination with metformin for the treatment duration of 26 weeks.
  Arms: Insulin degludec

SUMMARY:
This trial is conducted in Asia. The aim of this trial is to confirm the superiority of insulin degludec/liraglutide versus insulin degludec in controlling glycaemia in Chinese subjects with type 2 diabetes mellitus after 26 weeks of treatment

ELIGIBILITY:
Inclusion Criteria: Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including procedures to determine suitability for the trial - Male or female, age at least 18 years at the time of signing inform consent - Type 2 diabetes mellitus (clinically diagnosed) - HbA1c (glycosylated haemoglobin) above or equal to 7.5% by central laboratory analysis, with the aim of a median of 8.5%. When approximately 50% of the randomised subjects have an HbA1c above 8.5%, the remaining subjects randomised must have an HbA1c below or equal to 8.5% or when approximately 50% of the subjects randomised have an HbA1c below or equal to 8.5%, the remaining subjects randomised must have an HbA1c above 8.5% - Current treatment for at least 90 calendar days prior to screening with basal insulin plus metformin plus/minus α-glucosidase inhibitors, sulphonylureas, glinides or thiazolidinediones. Subjects should be on a stable dose for at least 60 calendar days prior to screening of: Basal insulin 20-50 units (U)/day (both inclusive) ( Individual fluctuations of plus/minus 5U during the 60 day period prior to the day of screening are acceptable.) on the day of screening in combination with: - Metformin (above or equal to 1500 mg or max tolerated dose) or - Metformin (above or equal to 1500 mg or max tolerated dose) and sulphonylureas (above or equal to half of the max approved dose according to local label) or - Metformin (above or equal to 1500 mg or max tolerated dose) and glinide (at least half of the max approved dose according to local label) or - Metformin (above or equal to 1500 mg or max tolerated dose) and α-glucosidase inhibitors (AGI) (at least half of the max approved dose according to local label) or - Metformin (above or equal to 1500 mg or max tolerated dose) and thiazolidinediones (at least half of the max approved dose according to local label) - Body mass index (BMI) above or equal to 24 kg/m^2 Exclusion Criteria: Current use of any antidiabetic drug (except for basal insulin, metformin, α-glucosidase inhibitors, sulphonylureas, glinides or thiazolidinediones) or anticipated change in concomitant medication, that in the investigator´s opinion could interfere with glucose level (e.g. systemic corticosteroids) - Treatment with glucagon like peptide -1 receptor agonists, or dipeptidyl-peptidase-4 inhibitors or insulin (except for basal insulin) within 90 days prior to Visit 1 - Impaired liver function defined as alanine aminotransferase above or equal to 2.5 times upper normal range - Impaired renal function defined as serum-creatinine above or equal to 133 μmol/L for males and above or equal to 125 μmol/L for females, or as defined according to local contraindications for metformin Screening calcitonin above or equal to 50 ng/L - Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia type 2 (MEN2) - Cardiac disorder defined as: congestive heart failure (NYHA class III-IV), diagnosis of unstable angina pectoris, cerebral stroke and/or myocardial infarction within the last 12 months prior to screening and/or planned coronary, carotid or peripheral artery revascularisation procedures - Severe uncontrolled treated or untreated hypertension (systolic blood pressure above or equal to 180 mm Hg or diastolic blood pressure above or equal to 100 mm Hg) - Proliferative retinopathy or maculopathy (macular oedema) requiring acute treatment - History of pancreatitis (acute or chronic)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 453 (Actual)
Dates: Start 2017-05-26 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2019-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR,1452), Study Director — Novo Nordisk A/S
Locations (25):
- China (24):
  - Novo Nordisk Investigational Site, Hefei, Anhui
  - Novo Nordisk Investigational Site, Beijing, Beijing Municipality
  - Novo Nordisk Investigational Site, Chongqing, Chongqing Municipality
  - Novo Nordisk Investigational Site, Fuzhou, Fujian
  - Novo Nordisk Investigational Site, Guangzhou, Guangdong
  - Novo Nordisk Investigational Site, Hengshui, Hebei
  - Novo Nordisk Investigational Site, Shijiazhuang, Hebei
  - Novo Nordisk Investigational Site, Tangshan, Hebei
  - Novo Nordisk Investigational Site, Harbin, Heilongjiang
  - Novo Nordisk Investigational Site, Yueyang, Hunan
  - Novo Nordisk Investigational Site, Hohhot, Inner Mongolia
  - Novo Nordisk Investigational Site, Changzhou, Jiangsu
  - Novo Nordisk Investigational Site, Nanjing, Jiangsu
  - Novo Nordisk Investigational Site, Zhenjiang, Jiangsu
  - Novo Nordisk Investigational Site, Nanchang, Jiangxi
  - Novo Nordisk Investigational Site, Changchun, Jilin
  - Novo Nordisk Investigational Site, Siping, Jilin
  - Novo Nordisk Investigational Site, Dalian, Liaoning
  - Novo Nordisk Investigational Site, Yinchuan, Ningxia
  - Novo Nordisk Investigational Site, Xi'an, Shaanxi
  - Novo Nordisk Investigational Site, Shanghai, Shanghai Municipality
  - Novo Nordisk Investigational Site, Taiyuan, Shanxi
  - Novo Nordisk Investigational Site, Tianjin, Tianjin Municipality
  - Novo Nordisk Investigational Site, Kunming, Yunnan
- Novo Nordisk Investigational Site, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 40 sites in China.
Pre-assignment Details: Participants were randomised in a 2:1 manner to receive either IDegLira or IDeg in combination with metformin.
Groups:
- Insulin Degludec/Liraglutide: Participants were to receive Insulin degludec/liraglutide (IDegLira) subcutaneous injection once daily in combination with metformin for 26 weeks. Participants received 16 dose steps (16 units insulin degludec and 0.6 mg liraglutide) initially. The dose was then adjusted twice weekly based on pre-breakfast self-measured plasma glucose (SMPG) values. The maximum dose was 50 dose steps (50 units IDeg/1.8 mg liraglutide). One dose step corresponded to 1 unit insulin degludec per 0.036 mg liraglutide.
- Insulin Degludec: Participants were to receive Insulin degludec (IDeg) subcutaneous injection once daily in combination with metformin for 26 weeks. Participants received 16 units insulin degludec initially. The dose was then adjusted twice weekly based on pre-breakfast SMPG values. The maximum dose was 50 units IDeg.
Period: Overall Study
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Started | 302 | 151
Treated | 301 | 151
Full Analysis Set (FAS) (FAS included all randomised participants.) | 302 | 151
Safety Analysis Set (SAS) (SAS included all participants who received at least one dose of IDegLira or IDeg.) | 301 | 151
Completed | 290 | 139
Not Completed | 12 | 12
Not completed — Adverse Event | 2 | 2
Not completed — Protocol Violation | 5 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Other | 2 | 3

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomised participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec | Total
Number analyzed (Participants) | 302 | 151 | 453
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.5 (9.8) | 55.3 (10.0) | 54.7 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 60 | 179
  Male | 183 | 91 | 274
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 302 | 151 | 453
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 302 | 151 | 453
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percentage of HbA1c] | 8.93 (1.20) | 8.96 (1.17) | 8.94 (1.19)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c
Description: Change in glycosylated haemoglobin (HbA1c) from baseline (week 0) to week 26 is presented.
Time Frame: Week 0, week 26
Population: FAS included all randomised participants. Overall number of participants analysed = participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage point of HbA1c
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 289 | 138
Percentage point of HbA1c | -1.93 (1.14) | -1.06 (1.19)
Statistical Analysis 1: Comparison: Insulin Degludec/Liraglutide vs Insulin Degludec; The response and change from baseline in response after 26 weeks are analysed using an analysis of covariance (ANCOVA) model with treatment and previous anti-diabetic treatment as fixed factors and corresponding baseline value as covariate; Test type: Superiority; p < .0001, ANCOVA; Treatment contrast = -0.92, 95% CI 2-sided [-1.09 to -0.75]

2. Secondary Outcome: Change in Body Weight
Description: Change in body weight from baseline (week 0) to week 26 is presented.
Time Frame: Week 0, week 26
Population: FAS included all randomised participants. Overall number of participants analysed = participants with available data.
Measure: Mean (Standard Deviation); unit: Kilogram (kg)
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 288 | 139
Kilogram (kg) | -0.7 (3.0) | 0.5 (2.7)

3. Secondary Outcome: Number of Treatment-emergent Severe or Blood Glucose (BG) Confirmed Hypoglycaemic Episodes
Description: Severe or BG confirmed hypoglycaemic episodes were defined as episodes that were severe according to the American Diabetes Association (ADA) classification (requiring assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions) or BG confirmed by a plasma glucose value < 3.1 millimoles per liter (mmol/L) with or without symptoms consistent with hypoglycaemia. Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product. Number of treatment-emergent severe or BG confirmed hypoglycaemic episodes during 26 weeks of treatment is presented.
Time Frame: Up to 26 weeks
Population: Safety analysis set (SAS) included all participants who received at least one dose of IDegLira or IDeg.
Measure: Number; unit: Episodes
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 301 | 151
Episodes | 38 | 36

4. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Change in FPG from baseline (week 0) to week 26 is presented.
Time Frame: Week 0, week 26
Population: FAS included all randomised participants. Overall number of participants analysed = participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 289 | 139
mmol/L | -3.57 (3.00) | -2.82 (3.15)

5. Secondary Outcome: Change in Waist Circumference
Description: Change in waist circumference from baseline (week 0) to week 26 is presented.
Time Frame: Week 0, week 26
Population: FAS included all randomised participants. Overall number of participants analysed = participants with available data.
Measure: Mean (Standard Deviation); unit: Centimeter (cm)
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 288 | 139
Centimeter (cm) | -0.4 (4.3) | 0.7 (3.3)

6. Secondary Outcome: Change in Mean of the 9-point Self-measured Plasma Glucose (SMPG) Profile
Description: Participants measured plasma glucose values using the blood glucose meter at 9 time points: before breakfast, 90 min after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 min after start of dinner, bedtime, at 4:00 am and before breakfast the following day. The mean of profile is defined as the area under the profile divided by measurement time and is calculated using the trapezoidal method. Change in mean of the 9-point SMPG profile from baseline (week 0) to week 26 is presented.
Time Frame: Week 0, week 26
Population: FAS included all randomised participants. Overall number of participants analysed = participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 272 | 133
mmol/L | -3.35 (2.63) | -2.31 (2.61)

7. Secondary Outcome: Change in SMPG-mean Post Prandial Increments
Description: Participants measured plasma glucose values using the blood glucose meter at 9 time points: before breakfast, 90 min after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 min after start of dinner, bedtime, at 4:00 am and before breakfast the following day. Change in SMPG-mean postprandial increment over all meals from baseline (week 0) to week 26 is presented.
Time Frame: Week 0, week 26
Population: FAS included all randomised participants. Overall number of participants analysed = participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 280 | 134
mmol/L | 0.08 (2.19) | 0.28 (2.71)

8. Secondary Outcome: Insulin Dose
Description: The mean of actual daily total insulin dose after 26 weeks of treatment is presented.
Time Frame: Week 26
Population: SAS included all participants who received at least one dose of IDegLira or IDeg. Overall number of participants analysed = participants with available data.
Measure: Mean (Standard Deviation); unit: Units of insulin (U)
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 290 | 139
Units of insulin (U) | 34.6 (11.1) | 37.9 (10.8)

9. Secondary Outcome: SMPG-9-point Profile (Individual Points in the Profile)
Description: Participants measured plasma glucose values using the blood glucose meter at 9 time points: before breakfast, 90 min after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 min after start of dinner, bedtime, at 4:00 am and before breakfast the following day. SMPG-9-point profile (individual points in the profile) at week 26 is presented.
Time Frame: Week 26
Population: FAS included all randomised participants. Number analysed = participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 302 | 151
mmol/L
  Before breakfast: number analyzed (Participants) | 282 | 136
  Before breakfast | 5.48 (1.06) | 5.88 (1.30)
  90 minutes after start of breakfast: number analyzed (Participants) | 279 | 131
  90 minutes after start of breakfast | 9.51 (2.66) | 10.50 (2.45)
  Before lunch: number analyzed (Participants) | 279 | 130
  Before lunch | 6.93 (2.10) | 8.17 (3.19)
  90 minutes after start of lunch: number analyzed (Participants) | 279 | 135
  90 minutes after start of lunch | 9.68 (2.52) | 11.21 (2.93)
  Before main evening meal: number analyzed (Participants) | 279 | 132
  Before main evening meal | 7.24 (2.16) | 7.87 (2.65)
  90 minutes after main evening meal: number analyzed (Participants) | 278 | 130
  90 minutes after main evening meal | 9.87 (2.53) | 10.86 (2.46)
  At bedtime: number analyzed (Participants) | 273 | 128
  At bedtime | 8.57 (2.52) | 9.52 (2.61)
  At 4:00 a.m.: number analyzed (Participants) | 270 | 131
  At 4:00 a.m. | 5.97 (1.49) | 6.61 (1.99)
  Before breakfast the following day: number analyzed (Participants) | 282 | 136
  Before breakfast the following day | 5.48 (1.14) | 5.83 (1.52)

10. Secondary Outcome: Change in Fasting High-density Lipoprotein (HDL) Cholesterol- Ratio to Baseline
Description: Change in fasting HDL cholesterol (measured in mmol/L) from baseline (week 0) to week 26 is presented as ratio to baseline.
Time Frame: Week 0, week 26
Population: FAS included all randomised participants. Overall number of participants analysed = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of HDL cholesterol
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 289 | 139
Ratio of HDL cholesterol | 1.00 (17.5) | 1.03 (15.9)

11. Secondary Outcome: Change in Fasting Low-density Lipoprotein (LDL) Cholesterol- Ratio to Baseline
Description: Change in fasting LDL cholesterol (measured in mmol/L) from baseline (week 0) to week 26 is presented as ratio to baseline.
Time Frame: Week 0, week 26
Population: FAS included all randomised participants. Overall number of participants analysed = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of LDL cholesterol
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 284 | 134
Ratio of LDL cholesterol | 0.89 (32.5) | 0.95 (37.7)

12. Secondary Outcome: Change in Fasting Very Low-density Lipoprotein (VLDL) Cholesterol- Ratio to Baseline
Description: Change in fasting VLDL cholesterol (measured in mmol/L) from baseline (week 0) to week 26 is presented as ratio to baseline.
Time Frame: Week 0, week 26
Population: FAS included all randomised participants. Overall number of participants analysed = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of VLDL cholesterol
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 289 | 139
Ratio of VLDL cholesterol | 0.92 (55.2) | 0.93 (49.1)

13. Secondary Outcome: Change in Fasting Total Cholesterol- Ratio to Baseline
Description: Change in fasting total cholesterol (measured in mmol/L) from baseline (week 0) to week 26 is presented as ratio to baseline.
Time Frame: Week 0, week 26
Population: FAS included all randomised participants. Overall number of participants analysed = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of total cholesterol
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 289 | 139
Ratio of total cholesterol | 0.92 (19.1) | 0.97 (20.0)

14. Secondary Outcome: Change in Fasting Triglycerides- Ratio to Baseline
Description: Change in fasting triglycerides (measured in mmol/L) from baseline (week 0) to week 26 is presented as ratio to baseline.
Time Frame: Week 0, week 26
Population: FAS included all randomised participants. Overall number of participants analysed = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of triglycerides
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 289 | 139
Ratio of triglycerides | 0.91 (63.7) | 0.92 (55.8)

15. Secondary Outcome: Change in Fasting Free Fatty Acids- Ratio to Baseline
Description: Change in fasting free fatty acids (measured in mmol/L) from baseline (week 0) to week 26 is presented as ratio to baseline.
Time Frame: Week 0, week 26
Population: FAS included all randomised participants. Overall number of participants analysed = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of free fatty acids
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 289 | 138
Ratio of free fatty acids | 0.65 (76.4) | 0.64 (61.9)

16. Secondary Outcome: Change in Fasting C-peptide- Ratio to Baseline
Description: Change in fasting C-peptide (measured in nanomoles per liter (nmol/L)) from baseline (week 0) to week 26 is presented as ratio to baseline.
Time Frame: Week 0, week 26
Population: FAS included all randomised participants. Overall number of participants analysed = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of C-peptide
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 286 | 137
Ratio of C-peptide | 0.64 (71.2) | 0.52 (71.8)

17. Secondary Outcome: Change in Fasting Insulin- Ratio to Baseline
Description: Change in fasting insulin (measured in picomoles per liter (pmol/L)) from baseline (week 0) to week 26 is presented as ratio to baseline.
Time Frame: Week 0, week 26
Population: FAS included all randomised participants. Overall number of participants analysed = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of insulin
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 288 | 139
Ratio of insulin | 0.63 (118.3) | 0.50 (106.4)

18. Secondary Outcome: Change in Fasting Glucagon- Ratio to Baseline
Description: Change in fasting glucagon (measured in picograms per milliliter (pg/mL)) from baseline (week 0) to week 26 is presented as ratio to baseline.
Time Frame: Week 0, week 26
Population: FAS included all randomised participants. Overall number of participants analysed = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of glucagon
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 287 | 138
Ratio of glucagon | 1.01 (95.8) | 1.09 (81.7)

19. Secondary Outcome: Change in HOMA-B (Beta-cell Function)- Ratio to Baseline
Description: Change in HOMA-B from baseline (week 0) to week 26 is presented as ratio to baseline.
Time Frame: Week 0, week 26
Population: FAS included all randomised participants. Overall number of participants analysed = participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio of beta-cell function
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 287 | 139
Ratio of beta-cell function | 1.47 (115.0) | 0.99 (113.4)

20. Secondary Outcome: Participants Who Achieved HbA1c < 7.0%, ADA Target (Yes/no)
Description: Participants who achieved HbA1c < 7.0%, ADA target (yes/no) is presented.
Time Frame: Week 26
Population: FAS included all randomised participants. Overall number of participants analysed = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 289 | 138
Participants
  Yes | 151 | 23
  No | 138 | 115

21. Secondary Outcome: Participants Who Achieved HbA1c ≤ 6.5%, American Association of Clinical Endocrinologists (AACE) Target (Yes/no)
Description: Participants who achieved HbA1c ≤ 6.5%, AACE target (yes/no) is presented.
Time Frame: Week 26
Population: FAS included all randomised participants. Overall number of participants analysed = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 289 | 138
Participants
  Yes | 96 | 10
  No | 193 | 128

22. Secondary Outcome: Participants Who Achieved HbA1c < 7.0% and Change From Baseline in Body Weight Below or Equal to Zero
Description: Participants who achieved HbA1c < 7.0% and change from baseline in body weight below or equal to zero is presented.
Time Frame: Week 26
Population: FAS included all randomised participants. Overall number of participants analysed = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 302 | 151
Participants
  Yes | 98 | 7
  No | 204 | 144

23. Secondary Outcome: Participants Who Achieved HbA1c ≤ 6.5% and Change From Baseline in Body Weight Below or Equal to Zero
Description: Participants who achieved HbA1c ≤ 6.5% and change from baseline in body weight below or equal to zero is presented.
Time Frame: Week 26
Population: FAS included all randomised participants. Overall number of participants analysed = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 302 | 151
Participants
  Yes | 59 | 3
  No | 243 | 148

24. Secondary Outcome: Participants Who Achieved HbA1c < 7.0% Without Treatment-emergent Severe or BG Confirmed Hypoglycaemic Episodes
Description: Severe or BG confirmed hypoglycaemic episodes were defined as episodes that were severe according to the ADA classification (required assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions) or BG confirmed by a plasma glucose value < 3.1 mmol/L with or without symptoms consistent with hypoglycaemia. Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product. Participants who achieved HbA1c < 7.0% at week 26 without treatment-emergent severe or BG confirmed hypoglycaemic episodes during the last 12 weeks of treatment is presented.
Time Frame: Week 26
Population: FAS included all randomised participants. Overall number of participants analysed = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 302 | 151
Participants
  Yes | 148 | 22
  No | 154 | 129

25. Secondary Outcome: Participants Who Achieved HbA1c ≤ 6.5% Without Treatment-emergent Severe or BG Confirmed Hypoglycaemic Episodes
Description: Severe or BG confirmed hypoglycaemic episodes were defined as episodes that were severe according to the ADA classification (required assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions) or BG confirmed by a plasma glucose value < 3.1 mmol/L with or without symptoms consistent with hypoglycaemia. Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product. Participants who achieved HbA1c ≤ 6.5% at week 26 without treatment-emergent severe or BG confirmed hypoglycaemic episodes during the last 12 weeks of treatment is presented.
Time Frame: Week 26
Population: FAS included all randomised participants. Overall number of participants analysed = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 302 | 151
Participants
  Yes | 93 | 9
  No | 209 | 142

26. Secondary Outcome: Participants Who Achieved HbA1c < 7.0% and Change From Baseline in Body Weight Below or Equal to Zero and Without Treatment-emergent Severe or BG Confirmed Hypoglycaemic Episodes
Description: Severe or BG confirmed hypoglycaemic episodes were defined as episodes that were severe according to the ADA classification (required assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions) or BG confirmed by a plasma glucose value < 3.1 mmol/L with or without symptoms consistent with hypoglycaemia. Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product. Participants who achieved HbA1c < 7.0% and change from baseline in body weight below or equal to zero and without treatment-emergent severe or BG confirmed hypoglycaemic episodes during the last 12 weeks of treatment is presented.
Time Frame: Week 26
Population: FAS included all randomised participants. Overall number of participants analysed = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 302 | 151
Participants
  Yes | 94 | 7
  No | 208 | 144

27. Secondary Outcome: Participants Who Achieved HbA1c ≤ 6.5% and Change From Baseline in Body Weight Below or Equal to Zero and Without Treatment-emergent Severe or BG Confirmed Hypoglycaemic Episodes
Description: Severe or BG confirmed hypoglycaemic episodes were defined as episodes that were severe according to the ADA classification (required assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions) or BG confirmed by a plasma glucose value < 3.1 mmol/L with or without symptoms consistent with hypoglycaemia. Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product. Participants who achieved HbA1c ≤ 6.5% and change from baseline in body weight below or equal to zero and without treatment-emergent severe or BG confirmed hypoglycaemic episodes during the last 12 weeks of treatment is presented.
Time Frame: Week 26
Population: FAS included all randomised participants. Overall number of participants analysed = participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 302 | 151
Participants
  Yes | 58 | 3
  No | 244 | 148

28. Secondary Outcome: Number of Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE was defined as an adverse event with onset date on or after the first day of exposure to randomised treatment and no later than seven days after the last day of randomised treatment. If the event had onset date before the first day of exposure on randomised treatment and increased in severity during the treatment period and until 7 days after the last drug date, then this event was considered as a TEAE.
Time Frame: Weeks 0-27
Population: SAS included all participants who received at least one dose of IDegLira or IDeg.
Measure: Number; unit: Adverse events
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 301 | 151
Adverse events | 641 | 230

29. Secondary Outcome: Number of Treatment-emergent Nocturnal Severe or BG Confirmed Hypoglycaemic Episodes
Description: Severe or BG confirmed hypoglycaemic episodes were defined as episodes that were severe according to the ADA classification (required assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions) or BG confirmed by a plasma glucose value < 3.1 mmol/L with or without symptoms consistent with hypoglycaemia. Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product. Nocturnal hypoglycaemic episodes were episodes occurring between 00:01 and 05.59 a.m. both inclusive. Number of treatment-emergent nocturnal severe or BG confirmed hypoglycaemic episodes is presented.
Time Frame: Weeks 0-27
Population: SAS included all participants who received at least one dose of IDegLira or IDeg.
Measure: Number; unit: Episodes
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 301 | 151
Episodes | 9 | 8

30. Secondary Outcome: Number of Treatment-emergent Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes
Description: Severe or BG confirmed hypoglycaemic episodes were defined as episodes that were severe according to the ADA classification (required assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions) or BG confirmed by a plasma glucose value < 3.1 mmol/L with symptoms consistent with hypoglycaemia. Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product. Number of treatment-emergent severe or BG confirmed symptomatic hypoglycaemic episodes is presented.
Time Frame: Weeks 0-27
Population: SAS included all participants who received at least one dose of IDegLira or IDeg.
Measure: Number; unit: Episodes
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 301 | 151
Episodes | 23 | 21

31. Secondary Outcome: Number of Treatment-emergent Nocturnal Severe or BG Confirmed Symptomatic Hypoglycaemic Episodes
Description: Severe or BG confirmed hypoglycaemic episodes were defined as episodes that were severe according to the ADA classification (required assistance of another person to actively administer carbohydrate, glucagon, or take other corrective actions) or BG confirmed by a plasma glucose value < 3.1 mmol/L with symptoms consistent with hypoglycaemia. Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product. Nocturnal hypoglycaemic episodes were episodes occurring between 00:01 and 05.59 a.m. both inclusive. Number of treatment-emergent nocturnal severe or BG confirmed symptomatic hypoglycaemic episodes is presented.
Time Frame: Weeks 0-27
Population: SAS included all participants who received at least one dose of IDegLira or IDeg.
Measure: Number; unit: Episodes
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 301 | 151
Episodes | 7 | 7

32. Secondary Outcome: Number of Treatment-emergent Hypoglycaemic Episodes According to ADA Definition
Description: Hypoglycaemic episodes were defined as treatment-emergent if the onset of the episode occurred on or after the first day of trial product administration, and no later than 7 calendar days after the last day on trial product. Number of treatment-emergent hypoglycaemic episodes according to ADA definition is presented.
Time Frame: Weeks 0-27
Population: SAS included all participants who received at least one dose of IDegLira or IDeg.
Measure: Number; unit: Episodes
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 301 | 151
Episodes | 1099 | 680

33. Secondary Outcome: Change in Physical Examination
Description: Physical examination parameters are categorised as cardiovascular system; central and peripheral nervous system; gastrointestinal system including mouth; general appearance; head, ears, eyes, nose, throat, neck; lymph node palpation; musculoskeletal system; respiratory system; skin and thyroid gland. The number of participants assessed as normal, abnormal not clinically significant (NCS) and abnormal clinically significant (CS) at week -2 and week 26 is presented.
Time Frame: Week -2, week 26
Population: SAS included all participants who received at least one dose of IDegLira or IDeg. "Number analyzed"=participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 301 | 151
Participants
  Week-2: Cardiovascular system: Normal | 299 | 149
  Week-2: Cardiovascular system: Abnormal NCS | 1 | 0
  Week-2: Cardiovascular system: Abnormal CS | 1 | 2
  Week 26: Cardiovascular system: number analyzed (Participants) | 288 | 139
  Week 26: Cardiovascular system: Normal | 286 | 137
  Week 26: Cardiovascular system: Abnormal NCS | 1 | 0
  Week 26: Cardiovascular system: Abnormal CS | 1 | 2
  Week-2: Central and peripheral nervous system: Normal | 299 | 150
  Week-2: Central and peripheral nervous system: Abnormal NCS | 2 | 0
  Week-2: Central and peripheral nervous system: Abnormal CS | 0 | 1
  Week 26: Central and peripheral nervous system: number analyzed (Participants) | 288 | 139
  Week 26: Central and peripheral nervous system: Normal | 287 | 139
  Week 26: Central and peripheral nervous system: Abnormal NCS | 1 | 0
  Week 26: Central and peripheral nervous system: Abnormal CS | 0 | 0
  Week -2: Gastrointestinal system: Normal | 299 | 150
  Week -2: Gastrointestinal system: Abnormal NCS | 2 | 1
  Week -2: Gastrointestinal system: Abnormal CS | 0 | 0
  Week 26: Gastrointestinal system: number analyzed (Participants) | 288 | 139
  Week 26: Gastrointestinal system: Normal | 285 | 139
  Week 26: Gastrointestinal system: Abnormal NCS | 2 | 0
  Week 26: Gastrointestinal system: Abnormal CS | 1 | 0
  Week -2: General appearance: Normal | 283 | 141
  Week -2: General appearance: Abnormal NCS | 11 | 2
  Week -2: General appearance: Abnormal CS | 7 | 8
  Week 26: General appearance: number analyzed (Participants) | 288 | 139
  Week 26: General appearance: Normal | 273 | 130
  Week 26: General appearance: Abnormal NCS | 9 | 2
  Week 26: General appearance: Abnormal CS | 6 | 7
  Week -2: Head, eyes, ENTand Neck: Normal | 295 | 147
  Week -2: Head, eyes, ENTand Neck: Abnormal NCS | 2 | 2
  Week -2: Head, eyes, ENTand Neck: Abnormal CS | 4 | 2
  Week 26: Head, eyes, ENTand Neck: number analyzed (Participants) | 288 | 139
  Week 26: Head, eyes, ENTand Neck: Normal | 283 | 137
  Week 26: Head, eyes, ENTand Neck: Abnormal NCS | 2 | 1
  Week 26: Head, eyes, ENTand Neck: Abnormal CS | 3 | 1
  Week -2: Lymph node palpation: Normal | 301 | 151
  Week -2: Lymph node palpation: Abnormal NCS | 0 | 0
  Week -2: Lymph node palpation: Abnormal CS | 0 | 0
  Week 26: Lymph node palpation: number analyzed (Participants) | 288 | 139
  Week 26: Lymph node palpation: Normal | 288 | 139
  Week 26: Lymph node palpation: Abnormal NCS | 0 | 0
  Week 26: Lymph node palpation: Abnormal CS | 0 | 0
  Week -2: Musculoskeletal system: Normal | 296 | 145
  Week -2: Musculoskeletal system: Abnormal NCS | 2 | 3
  Week -2: Musculoskeletal system: Abnormal CS | 3 | 3
  Week 26: Musculoskeletal system: number analyzed (Participants) | 288 | 139
  Week 26: Musculoskeletal system: Normal | 280 | 137
  Week 26: Musculoskeletal system: Abnormal NCS | 3 | 1
  Week 26: Musculoskeletal system: Abnormal CS | 5 | 1
  Week -2: Respiratory system: Normal | 301 | 151
  Week -2: Respiratory system: Abnormal NCS | 0 | 0
  Week -2: Respiratory system: Abnormal CS | 0 | 0
  Week 26: Respiratory system: number analyzed (Participants) | 288 | 139
  Week 26: Respiratory system: Normal | 288 | 139
  Week 26: Respiratory system: Abnormal NCS | 0 | 0
  Week 26: Respiratory system: Abnormal CS | 0 | 0
  Week -2: Skin: Normal | 270 | 132
  Week -2: Skin: Abnormal NCS | 22 | 13
  Week -2: Skin: Abnormal CS | 9 | 6
  Week 26: Skin: number analyzed (Participants) | 288 | 139
  Week 26: Skin: Normal | 259 | 126
  Week 26: Skin: Abnormal NCS | 22 | 9
  Week 26: Skin: Abnormal CS | 7 | 4
  Week -2: Thyroid gland: Normal | 295 | 147
  Week -2: Thyroid gland: Abnormal NCS | 4 | 2
  Week -2: Thyroid gland: Abnormal CS | 2 | 2
  Week 26: Thyroid gland: number analyzed (Participants) | 288 | 139
  Week 26: Thyroid gland: Normal | 284 | 134
  Week 26: Thyroid gland: Abnormal NCS | 3 | 3
  Week 26: Thyroid gland: Abnormal CS | 1 | 2

34. Secondary Outcome: Eye Examination
Description: Dilated fundoscopy or fundus photography was performed by the investigator at week -2 and week 26. The results of the examination were interpreted for each eye (left/right) are categorised as normal, abnormal NCS or abnormal CS. Number of participants in each category at week -2 and week 26 were presented.
Time Frame: Week -2, week 26
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 301 | 151
Participants
  Week -2: Left eye: Normal | 167 | 87
  Week -2: Left eye: Abnormal NCS | 34 | 15
  Week -2: Left eye: Abnormal CS | 100 | 49
  Week 26: Left eye: number analyzed (Participants) | 287 | 139
  Week 26: Left eye: Normal | 147 | 80
  Week 26: Left eye: Abnormal NCS | 35 | 14
  Week 26: Left eye: Abnormal CS | 105 | 45
  Week -2: Right eye: number analyzed (Participants) | 301 | 150
  Week -2: Right eye: Normal | 162 | 85
  Week -2: Right eye: Abnormal NCS | 41 | 18
  Week -2: Right eye: Abnormal CS | 98 | 47
  Week 26: Right eye: number analyzed (Participants) | 287 | 138
  Week 26: Right eye: Normal | 139 | 84
  Week 26: Right eye: Abnormal NCS | 37 | 12
  Week 26: Right eye: Abnormal CS | 111 | 42

35. Secondary Outcome: Change in Electrocardiogram (ECG)
Description: The ECG was assessed by the investigator at baseline (week -2) and week 26 and categorised as normal, abnormal NCS or abnormal CS. Number of participants in each ECG category at baseline and week 26 were presented.
Time Frame: Week -2, week 26
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 301 | 151
Participants
  Week -2: Normal | 175 | 90
  Week -2: Abnormal NCS | 76 | 41
  Week -2: Abnormal CS | 50 | 20
  Week 26: number analyzed (Participants) | 287 | 139
  Week 26: Normal | 175 | 91
  Week 26: Abnormal NCS | 73 | 32
  Week 26: Abnormal CS | 39 | 16

36. Secondary Outcome: Change in Pulse
Description: Change in pulse from baseline (week 0) to week 26 is presented.
Time Frame: Week 0, week 26
Population: SAS included all participants who received at least one dose of IDegLira or IDeg. Overall number of participants analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Beats per minute (beats/min)
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 288 | 139
Beats per minute (beats/min) | 5.7 (9.6) | 1.3 (8.7)

37. Secondary Outcome: Change in Blood Pressure (Systolic and Diastolic Blood Pressure)
Description: Change in blood pressure (systolic and diastolic blood pressure) from baseline (week 0) to week 26 is presented.
Time Frame: Week 0, week 26
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 288 | 139
Millimeters of mercury (mmHg)
  Systolic blood pressure | -3.5 (13.6) | -0.5 (12.5)
  Diastolic blood pressure | 0.1 (7.8) | -0.4 (8.1)

38. Secondary Outcome: Change in Biochemical Parameter- Amylase, Lipase, Creatinine Kinase, Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Alkaline Phosphatase (ALP)
Description: Change in amylase, lipase, creatinine kinase, ALT, AST, ALP from baseline (week 0) to week 26 is presented.
Time Frame: Week 0, week 26
Population: SAS included all participants who received at least one dose of IDegLira or IDeg. Number analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 289 | 139
Units per liter (U/L)
  Amylase | 10.45 (23.14) | 2.69 (11.72)
  Lipase | 16.97 (35.24) | -0.35 (13.81)
  Creatinine kinase | 3.32 (65.17) | 6.99 (84.31)
  ALT: number analyzed (Participants) | 288 | 139
  ALT | -3.02 (12.03) | -4.06 (11.97)
  AST: number analyzed (Participants) | 288 | 139
  AST | -1.42 (7.46) | -2.06 (7.92)
  ALP | -1.62 (13.30) | -1.70 (11.39)

39. Secondary Outcome: Change in Biochemical Parameter-calcium (Total), Albumin Corrected Calcium, Potassium, Sodium, Urea
Description: Change in calcium (total), albumin corrected calcium, potassium, sodium, urea from baseline (week 0) to week 26 is presented.
Time Frame: Week 0, week 26
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 289 | 139
mmol/L
  Calcium (total) | 0.01 (0.10) | -0.01 (0.09)
  Albumin corrected calcium: number analyzed (Participants) | 288 | 139
  Albumin corrected calcium | -0.00 (0.08) | -0.01 (0.08)
  Potassium | -0.03 (0.34) | -0.11 (0.35)
  Sodium | 1.03 (2.47) | 1.40 (2.43)
  Urea | -0.09 (1.32) | 0.17 (1.29)

40. Secondary Outcome: Change in Albumin
Description: Change in albumin from baseline (week 0) to week 26 is presented.
Time Frame: Week 0, week 26
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: Grams per deciliter (g/dL)
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 288 | 139
Grams per deciliter (g/dL) | 0.05 (0.29) | 0.02 (0.25)

41. Secondary Outcome: Change in Total Bilirubin
Description: Change in total bilirubin from baseline (week 0) to week 26 is presented.
Time Frame: Week 0, week 26
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 289 | 139
Micromoles per liter (umol/L) | -0.30 (3.89) | -0.54 (3.66)

42. Secondary Outcome: Change in Creatinine
Description: Change in creatinine from baseline (week 0) to week 26 is presented.
Time Frame: Week 0, week 26
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 289 | 139
umol/L | 0.44 (7.93) | -0.32 (7.52)

43. Secondary Outcome: Change in Total Protein
Description: Change in total protein from baseline (week 0) to week 26 is presented.
Time Frame: Week 0, week 26
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 289 | 139
g/dL | 0.08 (0.41) | 0.03 (0.39)

44. Secondary Outcome: Change in Haematological Parameter- Haematocrit
Description: Change in haematocrit from baseline (week 0) to week 26 is presented.
Time Frame: Week 0, week 26
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 289 | 139
Percentage of red blood cells | -0.07 (2.56) | -0.12 (2.14)

45. Secondary Outcome: Change in Haematological Parameter- Haemoglobin
Description: Change in haemoglobin from baseline (week 0) to week 26 is presented.
Time Frame: Week 0, week 26
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 288 | 139
mmol/L | -0.08 (0.52) | -0.09 (0.41)

46. Secondary Outcome: Change in Haematological Parameter- Leukocytes and Thrombocytes
Description: Change in leukocytes and thrombocytes from baseline (week 0) to week 26 is presented.
Time Frame: Week 0, week 26
Population: SAS included all participants who received at least one dose of IDegLira or IDeg. Number of participants analyzed = participants with available data.
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter (10^9/L)
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 289 | 138
10^9 cells per liter (10^9/L)
  Leukocytes | 0.32 (1.39) | 0.31 (1.18)
  Thrombocytes: number analyzed (Participants) | 287 | 138
  Thrombocytes | 14.13 (34.34) | 12.19 (34.01)

47. Secondary Outcome: Change in Haematological Parameter- Erythrocytes
Description: Change in erythrocytes from baseline (week 0) to week 26 is presented.
Time Frame: Week 0, week 26
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter (10^12/L)
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 289 | 139
10^12 cells per liter (10^12/L) | -0.06 (0.26) | -0.05 (0.24)

48. Secondary Outcome: Change in Haematological Parameter- Basophils
Description: Change in basophils from baseline (week 0) to week 26 is presented.
Time Frame: Week 0, week 26
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: Percentage of basophils
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 289 | 138
Percentage of basophils | 0.00 (0.34) | 0.01 (0.27)

49. Secondary Outcome: Change in Haematological Parameter- Eosinophils
Description: Change in eosinophils from baseline (week 0) to week 26 is presented.
Time Frame: Week 0, week 26
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: Percentage of eosinophils
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 289 | 138
Percentage of eosinophils | -0.15 (1.84) | -0.25 (1.72)

50. Secondary Outcome: Change in Haematological Parameter- Lymphocytes
Description: Change in lymphocytes from baseline (week 0) to week 26 is presented.
Time Frame: Week 0, week 26
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: Percentage of lymphocytes
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 289 | 138
Percentage of lymphocytes | -1.00 (6.95) | -0.82 (6.41)

51. Secondary Outcome: Change in Haematological Parameter- Monocytes
Description: Change in monocytes from baseline (week 0) to week 26 is presented.
Time Frame: Week 0, week 26
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: Percentage of monocytes
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 289 | 138
Percentage of monocytes | -0.19 (2.02) | -0.06 (2.19)

52. Secondary Outcome: Change in Haematological Parameter- Neutrophils
Description: Change in neutrophils from baseline (week 0) to week 26 is presented.
Time Frame: Week 0, week 26
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: Percentage of neutrophils
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 289 | 138
Percentage of neutrophils | 1.34 (7.85) | 0.99 (7.41)

53. Secondary Outcome: Change in Calcitonin
Description: Calcitonin levels were measured and were categorised as low, normal or high. Number of participants in each category at week 0 and week 26 were presented.
Time Frame: Week 0, week 26
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 301 | 151
Participants
  Week 0: Low | 0 | 0
  Week 0: Normal | 293 | 149
  Week 0: High | 8 | 2
  Week 26: number analyzed (Participants) | 289 | 139
  Week 26: Low | 0 | 0
  Week 26: Normal | 279 | 136
  Week 26: High | 10 | 3

54. Secondary Outcome: Urinalysis (Erythrocytes, Protein, Glucose and Ketones)
Description: The urinalysis was the measurements of protein, glucose, erythrocytes and ketones at week 0 and week 26 and categorised as negative, trace, 1+, 2+ and 3+. Number of participants in each category at week 0 and week 26 are presented.
Time Frame: Week 0, week 26
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 301 | 151
Participants
  Week 0: Erythrocytes: number analyzed (Participants) | 300 | 151
  Week 0: Erythrocytes: Negative | 258 | 121
  Week 0: Erythrocytes: Trace | 33 | 22
  Week 0: Erythrocytes: 1+ | 3 | 4
  Week 0: Erythrocytes: 2+ | 2 | 3
  Week 0: Erythrocytes: 3+ | 4 | 1
  Week 26: Erythrocytes: number analyzed (Participants) | 287 | 139
  Week 26: Erythrocytes: Negative | 255 | 120
  Week 26: Erythrocytes: Trace | 22 | 11
  Week 26: Erythrocytes: 1+ | 6 | 1
  Week 26: Erythrocytes: 2+ | 2 | 4
  Week 26: Erythrocytes: 3+ | 2 | 3
  Week 0: Glucose: number analyzed (Participants) | 300 | 151
  Week 0: Glucose: Negative | 171 | 92
  Week 0: Glucose: Trace | 33 | 13
  Week 0: Glucose: 1+ | 30 | 17
  Week 0: Glucose: 2+ | 25 | 13
  Week 0: Glucose: 3+ | 41 | 16
  Week 26: Glucose: number analyzed (Participants) | 287 | 139
  Week 26: Glucose: Negative | 256 | 110
  Week 26: Glucose: Trace | 14 | 16
  Week 26: Glucose: 1+ | 10 | 9
  Week 26: Glucose: 2+ | 4 | 2
  Week 26: Glucose: 3+ | 3 | 2
  Week 0: Ketones: number analyzed (Participants) | 300 | 151
  Week 0: Ketones: Negative | 274 | 137
  Week 0: Ketones: Trace | 21 | 10
  Week 0: Ketones: 1+ | 5 | 4
  Week 0: Ketones: 2+ | 0 | 0
  Week 0: Ketones: 3+ | 0 | 0
  Week 26: Ketones: number analyzed (Participants) | 287 | 139
  Week 26: Ketones: Negative | 272 | 132
  Week 26: Ketones: Trace | 14 | 7
  Week 26: Ketones: 1+ | 1 | 0
  Week 26: Ketones: 2+ | 0 | 0
  Week 26: Ketones: 3+ | 0 | 0
  Week 0: Protein: number analyzed (Participants) | 300 | 151
  Week 0: Protein: Negative | 172 | 89
  Week 0: Protein: Trace | 72 | 32
  Week 0: Protein: 1+ | 36 | 18
  Week 0: Protein: 2+ | 16 | 10
  Week 0: Protein: 3+ | 4 | 2
  Week 26: Protein: number analyzed (Participants) | 287 | 139
  Week 26: Protein: Negative | 198 | 89
  Week 26: Protein: Trace | 47 | 22
  Week 26: Protein: 1+ | 29 | 18
  Week 26: Protein: 2+ | 11 | 9
  Week 26: Protein: 3+ | 2 | 1

55. Secondary Outcome: Anti-insulin Degludec Specific Antibodies
Description: Serum samples were analysed for the presence of anti-insulin degludec specific antibodies. Results are presented as percentage of bound radioactivity-labelled insulin/total added radioactivity-labelled insulin (%B/T).
Time Frame: Week 27
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: %B/T
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 288 | 143
%B/T | 0.25 (1.25) | 0.13 (0.57)

56. Secondary Outcome: Antibodies Cross-reacting to Human Insulin
Description: Serum samples were analysed for the presence of antibodies cross-reacting to human insulin. Results are presented as percentage of bound radioactivity-labelled insulin/total added radioactivity-labelled insulin (%B/T).
Time Frame: Week 27
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: %B/T
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 288 | 143
%B/T | 9.07 (16.61) | 8.64 (16.84)

57. Secondary Outcome: Total Insulin Antibodies
Description: Serum samples were analysed for the presence of total insulin antibodies. Results are presented as percentage of bound radioactivity-labelled insulin/total added radioactivity-labelled insulin (%B/T).
Time Frame: Week 27
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: %B/T
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
Number analyzed (Participants) | 288 | 143
%B/T | 9.31 (17.33) | 8.77 (17.19)

58. Secondary Outcome: Occurrence of Anti-liraglutide Antibodies (Yes/no)
Description: This outcome measure is only applicable for the Insulin degludec/liraglutide treatment arm. Number of participants who measured with anti-liraglutide antibodies at week 27 are presented.
Time Frame: Week 27
Population: as for outcome 36
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide
Number analyzed (Participants) | 288
Participants
  Yes | 24
  No | 264

59. Secondary Outcome: Occurrence of Anti-liraglutide Antibodies Cross Reacting Native Glucagon-like Peptide-1 (GLP-1)
Description: This outcome measure is only applicable for the Insulin degludec/liraglutide treatment arm. Number of participants who measured with anti-liraglutide antibodies cross reacting native GLP-1 at week 27 are presented.
Time Frame: Week 27
Population: as for outcome 36
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide
Number analyzed (Participants) | 288
Participants
  Yes | 6

60. Secondary Outcome: Occurrence of Neutralising Liraglutide Antibodies
Description: This outcome measure is only applicable for the Insulin degludec/liraglutide treatment arm. Number of participants who measured with neutralising liraglutide antibodies at week 27 are presented.
Time Frame: Week 27
Population: as for outcome 36
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide
Number analyzed (Participants) | 288
Participants
  Yes | 0

61. Secondary Outcome: Occurrence of Neutralising Liraglutide Antibodies Cross Reacting Native GLP-1
Description: This outcome measure is only applicable for the Insulin degludec/liraglutide treatment arm. Number of participants who measured with neutralising liraglutide antibodies cross reacting native GLP-1 at week 27 are presented.
Time Frame: Week 27
Population: as for outcome 36
Measure: Count of Participants; unit: Participants
Arm/Group | Insulin Degludec/Liraglutide
Number analyzed (Participants) | 288
Participants
  Yes | 0

ADVERSE EVENTS:
Time Frame: Weeks 0-30
Description: All presented AEs are TEAEs. A TEAE was defined as an event that had onset date on or after the first day of exposure to trial product and no later than 7 days after the last day of trial product administration. Results are based on the SAS which included all participants who received at least one dose of IDegLira or IDeg.
Arm/Group | Insulin Degludec/Liraglutide | Insulin Degludec
All-Cause Mortality (participants affected / at risk) | 0/301 | 0/151
Serious Adverse Events (participants affected / at risk) | 13/301 | 7/151
Other Adverse Events (participants affected / at risk) | 113/301 | 43/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Degludec/Liraglutide (N=301) | Insulin Degludec (N=151)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Epiglottitis (Infections and infestations) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Thyroglossal cyst (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Degludec/Liraglutide (N=301) | Insulin Degludec (N=151)
Decreased appetite (Metabolism and nutrition disorders) | 21 (23) | 3 (3)
Diabetic retinopathy (Eye disorders) | 35 (35) | 11 (11)
Diarrhoea (Gastrointestinal disorders) | 22 (30) | 2 (2)
Lipase increased (Investigations) | 36 (38) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 38 (45) | 27 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-01-23): https://cdn.clinicaltrials.gov/large-docs/20/NCT03175120/SAP_000.pdf
  • Study Protocol (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/20/NCT03175120/Prot_001.pdf